CLINICAL TRIAL: NCT00468104
Title: Response to Instillation of Activase in the Pleural Cavity vs Placebo in the Management of Complicated Pleural Effusion/Empyema
Brief Title: Efficacy and Safety of Activase (Ateplase) vs Placebo in Complicated Pleural Effusions (CPE)/Empyemas
Acronym: CPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Pulmonary and Critical Care (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, GEORGE THOMMI, MD, Midwest Pulmonary and Critical Care
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11415
Record Dates: First submitted 2007-04-29; First posted 2007-05-02 (Estimated); Results first posted 2012-04-24 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Pleural Effusion Associated With Pulmonary Infection; Bacterial Pleural Effusion Other Than Tuberculosis
Keywords: parapneumonic pleural effusion; empyema; TPA (Activase, Alteplase)
MeSH Terms: conditions — Empyema | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alteplase, Placebo- intapleural instillation (Active Comparator): Either 25 mg of Alteplase or Placebo instilled daily. Response to therapy after three days. cross over to the other drug if no response was noted.
  Interventions: Drug: Alteplase; Drug: Placebo
- Placebo, Alteplase -2nd arm (Active Comparator): If the first arm fails then the 2nd arm ( cross over to either Placebo or Alteplase not used in the first arm) instilled intrapleurally daily for three days
  Interventions: Drug: Alteplase; Drug: Placebo

INTERVENTIONS:
Drug: Alteplase — 25 Mg of Alteplase in 100 cc of normal saline was instilled intrapeurally for daily for three days
Drug: Placebo — Placebo in 100 cc of normal saline was instilled intrapleurally daily for three days
  Other Names: TPA, Activase

SUMMARY:
The purpose of this study is to document the efficacy and safety of intrapleural instillation of Activase vs Placebo in the management of complicated pleural effusions and empyemas

DETAILED DESCRIPTION:
The current treatments available for complicated pleural effusions (CPE) include chest tube placement for drainage and IV antibiotics. If this fails and CPE occurs then in most patients thoracotomy is performed. Patients that are not surgical candidates have image guided catheter placement performed, sometimes multiple times. The American College of Chest Physicians (ACCP) formed a CPE panel and published guidelines for treating CPE. Percutaneous image-guided drainage is the most common approach for CPE. The panel recognizes the cumulative data that supports the use of fibrinolytics, VATS, and thoracotomy. The CPE panel acknowledged the lack of randomized clinical trials to determine efficacy and safety of these modalities in CPE and strongly encourages the research to take place.

Fibrinolytic therapy is a relatively noninvasive, easy to use, and is relatively inexpensive. If successful, it will prevent sepsis and septic shock, decrease hospital stay, morbidity and mortality and prevent any surgical procedures. Multiple doses of fibrinolytics have been used in CPE with no evidence of systemic anti-fibrinolytic activity. Complications with these medications are also very uncommon and only isolated instances are reported. The benefit from successful pleural drainage using these agents will decrease morbidity, mortality, surgical procedures, and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with complicated pleural effusions
* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age > 18 years

Exclusion Criteria

* Current use of oral anticoagulants (e.g., warfarin sodium) with an International Normalized Ratio (INR) >5- Activated partial thromboplastin time (aPPT) > 80, Platelet count < 100,000/mm3;
* Severe uncontrolled hypertension
* Recognized hypersensitivity to Activase; or any component of its formulation; Traumatic pleural effusion
* Pregnancy (positive pregnancy test)
* In another study for this condition
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation
* Recent stroke
* Intracranial hemorrhage
* arteriovenous malformation or aneurysm
* Intracranial neoplasm
* Acute myocardial infarction
* Acute pulmonary embolus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-04; Primary Completion 2008-10 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Thommi, MD, Principal Investigator — Midwest Pulmonary and Critical Care, PC
Locations (1):
- Nebraska Methodist Hospital, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with loculated pleural effusions that failed to respond to chest tube placement and standard medical treatment and were considered for surgery were given the option to enter into a double blind cross over trial
Pre-assignment Details: 108 patients were evaluated but only 100 entered the trial. 2 patients refused, 2 patients admitting physicians opted out of the trial, 3 patients chest tube removed inadvertently, 1 patient for coagulopathy
Groups:
- Alteplase Then Placebo: 25 mg of Alteplase in 100 cc of normal saline was instilled intrapleurally daily for three days. Chest CT scans were performed on the fourth day . If less than a 50% reduction in the pleural effusion was determined, the patient was given the option to go to surgery or to the second intervention of the trial (with Placebo)
- Placebo Then Alteplase: Placebo in 100 cc of normal saline was instilled intrapleurally daily for three days. Chest CT scans were performed on the fourth day . If less than a 50% reduction in the pleural effusion was determined, the patient was given the option to go to surgery or to the second intervention of the trial (with Alteplase)
Period: First Intervention
Arm/Group | Alteplase Then Placebo | Placebo Then Alteplase
Started | 54 | 46
Completed | 45 | 45
Not Completed | 9 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — bleeding at chest tube site--first dose | 1 | 0
Not completed — died within 3 weeks | 1 | 0
Not completed — malposition/blocked chest tube tube | 2 | 0
Not completed — large lung mass with minimal effusion | 1 | 0
Not completed — associated prolonged pneumothorax | 1 | 0
Not completed — trapped lung | 1 | 0
Period: Second Intervention
Arm/Group | Alteplase Then Placebo | Placebo Then Alteplase
Started | 8 (37 responded to Alteplase and did not go to the second intervention) | 41 (4 patients responded to Placebo and did not go to the second intervention)
Completed | 3 | 37
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 5 | 2
Not completed — discarded for malposition of chest tube | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Alteplase; Placebo: 25mg of Alteplase in 100 cc of normal saline instilled intrapleurally; 100 cc of normal saline instilled intrapleurally
Arm/Group | Alteplase; Placebo
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 67 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 64
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: No Surgical Intervention
Description: CT scans of the chest and Chest X rays (CXR) were used to determine resolution of Pleural effusions/empyema/ pneumonia after 3 days of Alteplase/ Placebo therapy. If no response was noted with the first intervention patients were offered surgery --Decortiation/ Video Assisted Thoracic Surgery (VATS) or to receive the second intervention. Patients that failed the second intervention were offered surgery.
Time Frame: patients were followed six weeks per protocol. Most patients treated with Alteplase were also followed for up to six months
Population: intention to treat
Measure: Number; unit: participants
Groups:
- Alteplase: 25mg of Alteplase in 100 cc of normal saline given intrapleurally daily for 3 days either in the first or second arm
- Placebo: Placebo in 100 cc of normal saline given daily intrapleurally for 3 days either in the first or second arm
Arm/Group | Alteplase | Placebo
Number analyzed (Participants) | 81 | 47
participants | 66 | 6
Statistical Analysis 1: Comparison: Alteplase vs Placebo; A univariate analysis was done to identify possible predictors of successful resolution of symptoms. The chi-square analysis was used to compare the percent successful; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Secondary Outcome: Number of Participants With Pneumonia That Responded to Therapy
Description: patients were followed for 6 weeks and CXR and CT scan were done to document resolution of pneumonia
Time Frame: 6 weeks
Population: protocol design prevented assigning symptom resolution to a specific intervention therefore secondary outcome measures in 6 weeks were not analyzed
Measure: Number; unit: participants
Groups:
- Alteplase: 25mg of Alteplase in 100 cc of normal saline instilled intrapleurally
- Placebo: 100 cc of normal saline instilled intrapleurally
Arm/Group | Alteplase | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Pleural Effusion/Empyema That Responded to Therapy
Description: patients were followed for 6 weeks and CXR and CT scan were done to document resolution of pleural effusion/empyema
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Alteplase | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Shortness of Breath That Responded to Therapy
Description: patients were followed for 6 weeks and clinical symptoms of resolution of shortness of breath were documented
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Alteplase | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Clinical Symptoms of Sepsis That Responded to Therapy
Description: patients were followed for 6 weeks and resolution of sepsis was documented
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Alteplase | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: soon after drug instillation and for the first 24 hours in the hospital and then followed up for six months
Description: adverse events that occurred in patients after they received both Alteplase and Placebo were placed in a separate group as we were unable to determine which intervention ( Alteplase or Placebo) caused the problem
Groups:
- Received Alteplase Only: These patients received only Alteplase and were not crossed over
- Received Placebo Only: These patients received Placebo only and were not crossed over
- Received Both Alteplase and Placebo: These patients were crossed over and received both Alteplase and Placebo
Arm/Group | Received Alteplase Only | Received Placebo Only | Received Both Alteplase and Placebo
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/8 | 0/40
Other Adverse Events (participants affected / at risk) | 10/42 | 5/8 | 8/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Received Alteplase Only (N=42) | Received Placebo Only (N=8) | Received Both Alteplase and Placebo (N=40)
serious bleeding at the chest tube site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — bleeding occurred soon after Alteplase instillation at the chest tube site--patient needed transfusion and was taken off the trial
Shortness of breath, worsening sepsis (General disorders) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Received Alteplase Only (N=42) | Received Placebo Only (N=8) | Received Both Alteplase and Placebo (N=40)
severe chest pain post drug instillation (General disorders) | 1 (12) | 0 (12) | 1 (12)
mild to moderate chest pain (General disorders) | 6 (12) | 1 (12) | 3 (12)
hypotension and worsening renal function (General disorders) | 0 (4) | 0 (4) | 4 (4) — congestive heart failure, cardiomyopathy and malignant pleural effusions patients had significant pleural fluid loss both with Alteplase and Placebo. These patients need careful fluid status and diuretics monitoring.
blood loss--pleural fluid (Blood and lymphatic system disorders) | 3 (3) | 0 (3) | 0 (3) — Patients effusion were bloody to start with and decreasing hemoglobin was noted over 2-3 days post drug instillation needing blood transfusion
increasing shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (2) — increasing SOB secondary to increasing pleural fluid
worsening sepsis (Infections and infestations) | 0 (2) | 2 (2) | 0 (2)

LIMITATIONS AND CAVEATS:
The sample size for secondary outcomes in the Placebo group is small

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No